CLINICAL TRIAL: NCT00085735
Title: A Study Evaluating Limited Target Volume Boost Irradiation and Reduced Dose Craniospinal Radiotherapy (18.00 Gy) and Chemotherapy in Children With Newly Diagnosed Standard Risk Medulloblastoma: A Phase III Double Randomized Trial
Brief Title: Comparison of Radiation Therapy Regimens in Combination With Chemotherapy in Treating Young Patients With Newly Diagnosed Standard-Risk Medulloblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0331; NCI-2009-00335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS0331; 12238; COG-ACNS0331; CDR0000365506; ACNS0331 (Other: Children's Oncology Group); ACNS0331 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2004-06-14; First posted 2004-06-16 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Craniospinal Irradiation; Cyclophosphamide; Lomustine; Radiotherapy; Radiation; Vincristine

ARMS (6):
- Arm I (3-7 years of age, LDCSI, IFRT) (Experimental): See Detailed Description (Arm I)
  Interventions: Drug: Cisplatin; Radiation: Craniospinal Irradiation; Drug: Cyclophosphamide; Radiation: Involved-Field Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Lomustine; Other: Quality-of-Life Assessment; Drug: Vincristine Sulfate
- Arm II (3-7 years of age, LDCSI, PFRT) (Experimental): See Detailed Description (Arm II)
  Interventions: Drug: Cisplatin; Radiation: Craniospinal Irradiation; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Lomustine; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Arm III (3-7 years of age, SDCSI, IFRT) (Experimental): See Detailed Description (Arm III)
  Interventions: Drug: Cisplatin; Radiation: Craniospinal Irradiation; Drug: Cyclophosphamide; Radiation: Involved-Field Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Lomustine; Other: Quality-of-Life Assessment; Drug: Vincristine Sulfate
- Arm IV (3-7 years of age, SDCSI, PFRT) (Active Comparator): See Detailed Description (Arm IV)
  Interventions: Radiation: Craniospinal Irradiation; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Lomustine; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Arm V (8-21 years of age, SDCSI, IFRT) (Experimental): See Detailed Description (Arm V)
  Interventions: Drug: Cisplatin; Radiation: Craniospinal Irradiation; Drug: Cyclophosphamide; Radiation: Involved-Field Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Lomustine; Other: Quality-of-Life Assessment; Drug: Vincristine Sulfate
- Arm VI (8-21 years of age, SDCSI, PFRT) (Active Comparator): See Detailed Description (Arm VI)
  Interventions: Drug: Cisplatin; Radiation: Craniospinal Irradiation; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Lomustine; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm I (3-7 years of age, LDCSI, IFRT); Arm II (3-7 years of age, LDCSI, PFRT); Arm III (3-7 years of age, SDCSI, IFRT); Arm V (8-21 years of age, SDCSI, IFRT); Arm VI (8-21 years of age, SDCSI, PFRT)
Radiation: Craniospinal Irradiation — Undergo craniospinal Irradiation
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Radiation: Involved-Field Radiation Therapy — Undergo smaller volume boost (involved-field radiation therapy)
  Other Names: IFRT; Involved field radiotherapy
  Arms: Arm I (3-7 years of age, LDCSI, IFRT); Arm III (3-7 years of age, SDCSI, IFRT); Arm V (8-21 years of age, SDCSI, IFRT)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lomustine — Given orally
  Other Names: 1-(2-Chloroethyl)-3-cyclohexyl-1-nitrosourea; 1-Nitrosourea, 1-(2-chloroethyl)-3-cyclohexyl-; Belustin; Belustine; CCNU; Cecenu; CeeNU; Chloroethylcyclohexylnitrosourea; Citostal; Gleostine; Lomeblastin; Lomustinum; Lucostin; Lucostine; N-(2-Chloroethyl)-N'-cyclohexyl-N-nitrosourea; Prava; RB-1509; WR-139017
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo standard volume boost (whole posterior fossa radiation therapy)
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm II (3-7 years of age, LDCSI, PFRT); Arm IV (3-7 years of age, SDCSI, PFRT); Arm VI (8-21 years of age, SDCSI, PFRT)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase III trial is studying how well standard-dose radiation therapy works compared to reduced-dose radiation therapy in children 3-7 years of age AND how well standard volume boost radiation therapy works compared to smaller volume boost radiation therapy when given together with chemotherapy in treating young patients who have undergone surgery for newly diagnosed standard-risk medulloblastoma. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as vincristine, cisplatin, lomustine, and cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving radiation therapy with chemotherapy after surgery may kill any remaining tumor cells. It is not yet known whether standard-dose radiation therapy is more effective than reduced-dose radiation therapy when given together with chemotherapy after surgery in treating young patients with medulloblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether reducing the craniospinal dose of radiation therapy to 18.00 Gy in children 3-7 years of age does not compromise event-free survival and overall survival as compared to treatment with 23.40 Gy of craniospinal radiation; and to determine if reducing the irradiated volume of the primary site tumor boost from the whole posterior fossa to the tumor bed only will not compromise event-free and overall survival.

SECONDARY OBJECTIVES:

I. To evaluate patterns of failure in children treated with an irradiation boost volume smaller than conventional posterior fossa volumes.

II. To reduce the cognitive, auditory and endocrinologic effects of treatment of average-risk medulloblastoma by reducing the dose of craniospinal irradiation therapy.

III. To determine if the audiologic and endocrinologic toxicity will be reduced with the use of limited tumor boost volume irradiation compared to patients treated with conventional target volumes of radiation.

IV. To develop an optimal gene expression medulloblastoma outcome predictor, validated prospectively in a multi-institution randomized clinical trial.

V. To improve compliance with long-term quality of life and functional status data submission by educating institutional nurses to administer and submit for analysis a battery of four instruments: Behavior Assessment System for Children- 2nd Edition (BASC-2), Adaptive Behavior Assessment System - 2nd Edition (ABAS-II), Behavior Rating Inventory of Executive Function (BRIEF), PedsQLTM 4.0.

OUTLINE: Patients 3-7 years of age are randomized to 1 of 4 arms (Arm I-IV). Patients 8-21 years of age are randomized to 1 of 2 arms (Arm V or VI).

Within 31 days after definitive surgery, all patients begin therapy. Patients undergo radiation therapy with doses according to their Arm randomization on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47 (weeks 0-6). All patients receive vincristine intravenously (IV) over 1 minute (or infusion via minibag as per institutional policy) on days 8, 15, 22, 29, 36, and 43 (weeks 1-6).

ARM I: Patients 3-7 years of age undergo lowered dose craniospinal irradiation (LDCSI) with involved-field radiation therapy (IFRT) boost.

ARM II: Patients 3-7 years of age undergo LDCSI with whole posterior fossa radiation therapy (PFRT) boost.

ARM III: Patients 3-7 years of age undergo standard dose craniospinal irradiation (SDCSI) with IFRT boost.

ARM IV: Patients 3-7 years of age undergo SDCSI with PFRT boost.

ARM V: Patients 8-21 years of age undergo SDCSI with IFRT boost.

ARM VI: Patients 8-21 years of age undergo SDCSI with PFRT boost.

MAINTENANCE CHEMOTHERAPY: Beginning 4 weeks after completion of chemoradiotherapy, patients receive 2 different regimens of maintenance chemotherapy for a total of 9 courses. Each course in regimen A is 6 weeks (42 days) in duration. Each course in regimen B is 4 weeks (28 days) in duration.

REGIMEN A (courses 1, 2, 4, 5, 7, and 8): Patients receive lomustine orally and cisplatin IV over 6 hours on day 1 and vincristine IV on days 1, 8, and 15 of weeks 11, 17, 27, 33, 43, and 49.

REGIMEN B (courses 3, 6, and 9): Patients receive cyclophosphamide IV over 1 hour on days 1 and 2 and vincristine IV on days 1 and 8 of weeks 23, 39, and 55.

Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at 3-6 months after completion of radiotherapy and at 3-4 years after study entry. Neurocognitive function may also be assessed.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

OUTLINE: Patients 3-7 years of age are randomized to 1 of 4 arms (Arm I-IV). Patients 8-21 years of age are randomized to 1 of 2 arms (Arm V or VI).

Within 31 days after definitive surgery, all patients begin therapy. Patients undergo radiation therapy with doses according to their Arm randomization on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47 (weeks 0-6). All patients receive vincristine intravenously (IV) over 1 minute (or infusion via minibag as per institutional policy) on days 8, 15, 22, 29, 36, and 43 (weeks 1-6).

ARM I: Patients 3-7 years of age undergo lowered dose craniospinal irradiation (LDCSI) with involved-field radiation therapy (IFRT) boost.

ARM II: Patients 3-7 years of age undergo LDCSI with whole posterior fossa radiation therapy (PFRT) boost.

ARM III: Patients 3-7 years of age undergo standard dose craniospinal irradiation (SDCSI) with IFRT boost.

ARM IV: Patients 3-7 years of age undergo SDCSI with PFRT boost.

ARM V: Patients 8-21 years of age undergo SDCSI with IFRT boost.

ARM VI: Patients 8-21 years of age undergo SDCSI with PFRT boost.

MAINTENANCE CHEMOTHERAPY: Beginning 4 weeks after completion of chemoradiotherapy, patients receive 2 different regimens of maintenance chemotherapy for a total of 9 courses. Each course in regimen A is 6 weeks (42 days) in duration. Each course in regimen B is 4 weeks (28 days) in duration.

REGIMEN A (courses 1, 2, 4, 5, 7, and 8): Patients receive lomustine orally and cisplatin IV over 6 hours on day 1 and vincristine IV on days 1, 8, and 15 of weeks 11, 17, 27, 33, 43, and 49.

REGIMEN B (courses 3, 6, and 9): Patients receive cyclophosphamide IV over 1 hour on days 1 and 2 and vincristine IV on days 1 and 8 of weeks 23, 39, and 55.

Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at 3-6 months after completion of radiotherapy and at 3-4 years after study entry. Neurocognitive function may also be assessed.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed medulloblastoma located in the posterior fossa

  * Standard-risk disease
* Minimal volume, non-disseminated disease, defined by the following:

  * Residual tumor ≤ 1.5 cm^2 confirmed by MRI with contrast imaging within 21 days after surgery
  * No metastatic disease in the head, spine, or cerebrospinal fluid (CSF) confirmed by both of the following:

    * Enhanced MRI of the spine within 5 days before surgery OR within 28 days after surgery
    * Negative cytological examination of CSF after surgery, but before study enrollment
* Brain stem involvement allowed
* Performance status - Karnofsky 50-100% (> 16 years of age)
* Performance status - Lansky 30-100% (≤ 16 years of age)
* Absolute neutrophil count > 1,500/uL
* Platelet count > 100,000/uL (transfusion independent)
* Hemoglobin > 10 g/dL (transfusions allowed)
* Bilirubin < 1.5 times upper limit of normal (ULN) for age
* AST or ALT < 1.5 times ULN for age
* Creatinine clearance OR radioisotope glomerular filtration rate >= 70 mL/min/1.73m^2 or a serum creatinine based on age/gender as follows:

Age Maximum Serum Creatine (mg/dL)

* 1month to < 6 months male: 0.4 female: 0.4
* 6 months to <1 year male: 0.5 female: 0.5
* 1 year to < 2 years male: 0.6 female: 0.6
* 2 to < 6 years male: 0.8 female: 0.8
* 6 to < 10 years male: 1 female: 1
* 10 to < 13 years male: 1.2 female: 1.2
* 13 to < 16 years male: 1.5 female: 1.4
* >= 16 years male: 1.7 female: 1.4

  * Not pregnant or nursing
  * Negative pregnancy test
  * Fertile patients must use effective contraception
  * No prior chemotherapy
  * Prior corticosteroids allowed
  * No prior radiotherapy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 549 (Actual)
Dates: Start 2004-04-30 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff M Michalski, Principal Investigator — Children's Oncology Group
Locations (197):
- United States (174):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Children's Hospital and Clinic-Saint Paul, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (14):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Dutch Childhood Oncology Group, Utrecht, Netherlands
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Switzerland (3):
  - Swiss Pediatric Oncology Group - Bern, Bern
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

REFERENCES:
- [Derived] Michalski JM, Janss AJ, Vezina LG, Smith KS, Billups CA, Burger PC, Embry LM, Cullen PL, Hardy KK, Pomeroy SL, Bass JK, Perkins SM, Merchant TE, Colte PD, Fitzgerald TJ, Booth TN, Cherlow JM, Muraszko KM, Hadley J, Kumar R, Han Y, Tarbell NJ, Fouladi M, Pollack IF, Packer RJ, Li Y, Gajjar A, Northcott PA. Children's Oncology Group Phase III Trial of Reduced-Dose and Reduced-Volume Radiotherapy With Chemotherapy for Newly Diagnosed Average-Risk Medulloblastoma. J Clin Oncol. 2021 Aug 20;39(24):2685-2697. doi: 10.1200/JCO.20.02730. Epub 2021 Jun 10. PMID 34110925
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants 3-21 years of age were recruited at Children's Oncology Group institutions worldwide and at sites affiliated with the Dutch Childhood Oncology Group. The first patient was enrolled on April 30, 2004 and the last patient was enrolled on January 6, 2014.
Pre-assignment Details: Patients were randomized to receive a smaller volume boost (radiation to tumor bed)(IFRT) or standard volume boost (radiation to the entire posterior fossa) (PFRT).Patients 3-7 years of age were also randomized to receive reduced-dose craniospinal radiation (LDCSI) or standard-dose craniospinal radiation (SDCSI).Patients 8 and older received SDCSI.
Groups:
- Arm I (3-7 Yrs of Age, LDCSI, IFRT): Patients 3-7 years of age, LDCSI, IFRT
- Arm II (3-7 Yrs of Age, LDCSI, PFRT): Patients 3-7 years of age, LDCSI, PFRT
- Arm III (3-7 Yrs of Age, SDCSI, IFRT): Patients 3-7 years of age, SDCSI, IFRT
- Arm IV (3-7 Yrs of Age, SDCSI, PFRT): Patients 3-7 years of age, SDCSI, PFRT
- Arm V (8-21 Yrs of Age, SDCSI, IFRT): Patients 8-21 years of age, SDCSI, IFRT
- Arm VI (8-21 Yrs of Age, SDCSI, PFRT): Patients 8-21 yrs of age, SDCSI, PFRT
Period: Overall Study
Arm/Group | Arm I (3-7 Yrs of Age, LDCSI, IFRT) | Arm II (3-7 Yrs of Age, LDCSI, PFRT) | Arm III (3-7 Yrs of Age, SDCSI, IFRT) | Arm IV (3-7 Yrs of Age, SDCSI, PFRT) | Arm V (8-21 Yrs of Age, SDCSI, IFRT) | Arm VI (8-21 Yrs of Age, SDCSI, PFRT)
Started | 64 | 64 | 63 | 65 | 147 | 146
Completed | 52 | 54 | 46 | 46 | 105 | 115
Not Completed | 12 | 10 | 17 | 19 | 42 | 31
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 4 | 6 | 3 | 4 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 3 | 2 | 3 | 11 | 8
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 5 | 7 | 8
Not completed — Patient ineligible | 1 | 0 | 3 | 7 | 17 | 8
Not completed — Excess residual disease | 2 | 2 | 1 | 1 | 1 | 4
Not completed — Reason not documented | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Pt transferred to inst w/out study open | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only eligible patients are included in each of the 6 groups for baseline characteristics.
Groups:
- Arm I (3-7 Years of Age, LDCSI, IFRT): Eligible patients 3-7 yrs of age, LDCSI, IFRT
- Arm II (3-7 Years of Age, LDCSI, PFRT): Eligible patients 3-7 yrs of age, LDCSI, PFRT
- Arm III (3-7 Years of Age, SDCSI, IFRT): Eligible patients 3-7 yrs of age, SDCSI, IFRT
- Arm IV (3-7 Years of Age, SDCSI, PFRT): Eligible patients 3-7 yrs of age, SDCSI, PFRT
- Arm V (8-21 Years of Age, SDCSI, IFRT): Eligible patients 8-21 yrs of age, SDCSI, IFRT
- Arm VI (8-21 Years of Age, SDCSI, PFRT): Eligible patients 8-21 yrs of age, SDCSI, PFRT
- Total: Total of all reporting groups
Arm/Group | Arm I (3-7 Years of Age, LDCSI, IFRT) | Arm II (3-7 Years of Age, LDCSI, PFRT) | Arm III (3-7 Years of Age, SDCSI, IFRT) | Arm IV (3-7 Years of Age, SDCSI, PFRT) | Arm V (8-21 Years of Age, SDCSI, IFRT) | Arm VI (8-21 Years of Age, SDCSI, PFRT) | Total
Number analyzed (Participants) | 63 | 64 | 60 | 58 | 130 | 138 | 513
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 63 | 64 | 60 | 58 | 120 | 128 | 493
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 10 | 10 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 5.9 [3.2 to 7.8] | 5.9 [3.3 to 7.9] | 5.9 [3.0 to 8.0] | 5.4 [3.1 to 7.7] | 12.4 [8.0 to 19.8] | 11.8 [8 to 21.8] | 8.3 [3.0 to 21.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 20 | 24 | 53 | 51 | 184
  Male | 47 | 44 | 40 | 34 | 77 | 87 | 329
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 8 | 9 | 19 | 23 | 87
  Not Hispanic or Latino | 51 | 44 | 50 | 46 | 110 | 109 | 410
  Unknown or Not Reported | 2 | 2 | 2 | 3 | 1 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 2 | 2 | 4 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 2 | 0 | 0 | 5
  Black or African American | 5 | 6 | 5 | 3 | 13 | 9 | 41
  White | 50 | 48 | 46 | 48 | 108 | 120 | 420
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 5 | 3 | 4 | 7 | 35

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time interval from date of study entry to date of disease progression, disease recurrence, second malignant neoplasm or death from any cause, whichever occurs first, or to the date of last follow-up for patients without events. EFS was estimated using the method of Kaplan and Meier. 3-year estimates are reported with 95% confidence intervals (CI's).
Time Frame: Assessed at 3 years
Population: Per protocol only eligible & evaluable pts are included. Pts with anaplastic histology or disseminated/excess residual disease were not evaluable (NE). 26/23 IFRT/PFRT pts were NE, leaving 227 vs 237 for this comparison. The LD/SD CSI comparison was done only in pts 3-7 yrs of age. 11/8 LD/SDCSI pts were NE, leaving 116 vs 110 for this comparison.
Measure: Number (95% Confidence Interval); unit: probability of 3 year EFS
Groups:
- Low-dose Craniospinal Radiation (LDSCI): Includes eligible patients 3-7 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the LDCSI arms (Arms I and II)
- Standard-dose Craniospinal Radiation (SDCSI): Includes eligible patients 3-7 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the SDCSI arms (Arms III and IV)
- Involved Field Radiation (IFRT): Includes eligible patients without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the IFRT arms (I, III, V).
- Posterior Fossa Radiation (PFRT): Includes eligible patients without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the PFRT arms (II, IV, VI).
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI) | Involved Field Radiation (IFRT) | Posterior Fossa Radiation (PFRT)
Number analyzed (Participants) | 116 | 110 | 227 | 237
probability of 3 year EFS
  LDCSI vs SDCSI: number analyzed (Participants) | 116 | 110 | 0 | 0
  LDCSI vs SDCSI | 76.3 [67.9 to 84.7] | 84.9 [77.6 to 92.2] |  |
  IFRT vs PFRT: number analyzed (Participants) | 0 | 0 | 227 | 237
  IFRT vs PFRT |  |  | 85.8 [81.1 to 90.5] | 85.8 [81.1 to 90.5]
Statistical Analysis 1: Comparison: Low-dose Craniospinal Radiation (LDSCI) vs Standard-dose Craniospinal Radiation (SDCSI); The comparison is based on all eligible randomized patients 3-7 years of age without anaplastic histology or excess residual disease or disseminated disease by central review per the protocol document. Using a one-sided log rank test with type I error of 0.20, this study was designed to have power of 0.80 to detect a 10% reduction in cure rate due to the use of LDCSI compared to SDCSI; Test type: Non-Inferiority — A hazard ratio of 1.6 is used as the non-inferiority margin. For the final analysis of comparing LDCSI vs. SDCSI, a one-sided 80% upper confidence limit of the hazard ratio based on a stratified approach will be estimated (stratified by RT group (IFRT vs. PFRT)). If the upper confidence limit is lower than 1.6, LDCSI would be deemed to be non-inferior. If not, non-inferiority would not be established; Hazard Ratio (HR) = 1.5, 80% CI 1-sided [upper limit 1.9]
Statistical Analysis 2: Comparison: Involved Field Radiation (IFRT) vs Posterior Fossa Radiation (PFRT); The comparison is based on all eligible randomized patients 3-21 years of age without anaplastic histology or excess residual disease or disseminated disease by central review as per the protocol document. Using a one-sided log rank test with type I error of 0.20, this study was designed with power of 0.94 to detect a 10% reduction in cure rate and power of 0.65 to detect a 5% reduction in cure rate, due to the use of IFRT compared to PFRT; Test type: Non-Inferiority — A hazard ratio of 1.6 is used as the non-inferiority margin. For the final analysis comparing IFRT vs. PFRT, a one-sided 94% upper confidence limit of the hazard ratio based on a stratified approach will be estimated (stratified by age group and RT group (LDCSI vs. SDCSI)). If the upper confidence limit is lower than 1.6, IFRT would be deemed to be non-inferior. If not, non-inferiority would not be established; Hazard Ratio (HR) = 1.0, 94% CI 1-sided [upper limit 1.3]

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from date of study entry to date of death from any cause or to the date of last follow-up for survivors. OS was estimated using the method of Kaplan and Meier. 3-year estimates are reported with 95% CI's. For purposes of this analysis, arms I, III and V (involved field radiation therapy [IFRT]) are combined and compared to arms II, IV and VI (posterior fossa irradiation [PFRT]).
Time Frame: 3 years
Population: Per protocol only eligible & evaluable pts were included.Pts with anaplastic histology or disseminated/excess residual disease were not evaluable (NE). 26/23 IFRT/PFRT pts were NE, leaving 227 vs 237 for this comparison. The LD/SD CSI comparison was done only in pts 3-7 yrs of age. 11/8 LD/SDCSI pts were NE, leaving 116 vs 110 for this comparison.
Measure: Number (95% Confidence Interval); unit: Probability of 3 yr OS rate
Groups:
- Low-dose Craniospinal Radiation (LDSCI): Includes eligible patients 3-7 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the LDCSI arms (Treatment Arms I or II)
- Standard-dose Craniospinal Radiation (SDCSI): Includes eligible patients 3-7 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the SDCSI arms (Treatment Arms III or IV)
- Involved Field Radiation (IFRT): Includes eligible patients 3-21 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the IFRT arms (Treatment Arms I, III, V)
- Posterior Fossa Radiation (PFRT): Includes eligible patients 3-21 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the PFRT arms (Treatment Arms II, IV, VI)
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI) | Involved Field Radiation (IFRT) | Posterior Fossa Radiation (PFRT)
Number analyzed (Participants) | 116 | 110 | 227 | 237
Probability of 3 yr OS rate
  IFRT vs PFRT: number analyzed (Participants) | 0 | 0 | 227 | 237
  IFRT vs PFRT |  |  | 90.3 [86.2 to 94.4] | 93.3 [90.0 to 96.6]
  LDCSI vs SDCSI: number analyzed (Participants) | 116 | 110 | 0 | 0
  LDCSI vs SDCSI | 85.5 [78.4 to 92.6] | 90.4 [84.3 to 96.5] |  |

3. Secondary Outcome: Local Posterior Fossa (LPF) Failure Rate
Description: LPF failure was defined as tumor recurrence/progression within the tumor bed. The cumulative incidence (CI) of LPF failure was estimated; 3-year estimates were reported with 95% confidence intervals. Patients with other failure types (e.g., NPF) and with other events prior to LPF failure (e.g., death, second malignancy) were considered as having competing events.
Time Frame: 3 years
Population: Eligible and evaluable patients 3-21 yrs of age are included. Patients with anaplastic histology or disseminated/excess residual disease were not evaluable (NE). Arms I/III/V [IFRT] are combined & arms II/IV/VI [PFRT] are combined. 26 & 23 IFRT & PFRT pts were NE and were excluded, leaving 227 and 237 eligible and evaluable pts.
Measure: Number (95% Confidence Interval); unit: percentage 3 yr cumulative incidence
Arm/Group | Involved Field Radiation (IFRT) | Posterior Fossa Radiation (PFRT)
Number analyzed (Participants) | 227 | 237
percentage 3 yr cumulative incidence | 1.4 [0.0 to 2.89] | 2.7 [0.6 to 4.9]

4. Secondary Outcome: Non-local Posterior Fossa (NLPF) Failure Rate
Description: NLPF failure was defined as tumor recurrence/progression outside the radiation therapy clinical target volume boost (CTV-boost) but within the posterior fossa CTV (CTV-PF). The cumulative incidence (CI) of NLPF failure was estimated; 3-year estimates were reported with 95% confidence intervals. Patients with other failure types (e.g., NPF, LPF) and with other events prior to NLPF failure (e.g., death, second malignancy) were considered as having competing events.
Time Frame: 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of 3 yr cumulative incidence
Arm/Group | Involved Field Radiation (IFRT) | Posterior Fossa Radiation (PFRT)
Number analyzed (Participants) | 227 | 237
Percentage of 3 yr cumulative incidence | 6.9 [3.5 to 10.3] | 2.7 [0.6 to 4.8]

5. Secondary Outcome: Non-posterior Fossa (NPF) Failure Rate
Description: NPF failure was defined as tumor recurrence within the neuroaxis but outside the radiation therapy clinical target volume (CTV). The cumulative incidence (CI) of NPF failure was estimated; 3-year estimates were reported with 95% confidence intervals. Patients with other failure types (e.g., LPF failure) and with other events prior to NPF failure (e.g., death, second malignancy) were considered as having competing events.
Time Frame: 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of 3 yr cumulative incidence
Arm/Group | Involved Field Radiation (IFRT) | Posterior Fossa Radiation (PFRT)
Number analyzed (Participants) | 227 | 237
Percentage of 3 yr cumulative incidence | 5.1 [2.2 to 8.0] | 6.2 [3.0 to 9.4]

6. Secondary Outcome: Post-treatment Endocrine Function by CSI Group
Description: Post-treatment endocrine function was measured by laboratory assessment of the thyroid stimulating hormone (TSH). The mean TSH will be reported.
Time Frame: Up to 3 years
Population: Only eligible & evaluable pts 3-7 years of age were included. Pts with anaplastic histology or disseminated/excess residual disease were not evaluable (NE). 11 and 8 LDSCI and SDCSI pts were NE, respectively, leaving 116 vs 110 for this comparison. Of these, 89 LDSCI and 79 SDCSI pts had post-treatment TSH values available and were included.
Measure: Mean (Standard Deviation); unit: uU/ml
Groups:
- Low-dose Craniospinal Radiation (LDSCI): Includes eligible patients 3-7 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the LDCSI arms (Treatment Arms I or II) and with a post-treatment TSH value.
- Standard-dose Craniospinal Radiation (SDCSI): Includes eligible patients 3-7 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and randomized to one of the SDCSI arms (Treatment Arms III or IV) and with a post-treatment TSH value.
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 89 | 79
uU/ml | 5.3 (5.6) | 6.1 (5.3)

7. Secondary Outcome: Post-treatment Grade 3+ Hearing Loss as Measured by Common Terminology Criteria for Adverse Events (CTCAE) Version (v)4
Description: Proportions of patients with grade 3+ hearing loss after the completion of therapy will be calculated and reported separately for low dose craniospinal irradiation (LDCSI) versus (vs.) standard dose craniospinal irradiation (SDCSI) patients. Eligible and evaluable patients 3-7 years of age will be used.
Time Frame: Up to 3 years
Population: Only eligible & evaluable pts 3-7 years of age are included since only younger pts were randomized to either LD or SD CSI. 11 and 8 LDCSI and SDCSI pts respectively were not evaluable due to anaplastic disease or excess residual/disseminated disease, leaving 116 vs 110 patients for this analysis.
Measure: Number; unit: Percentage of pts with g3+ hearing loss
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 116 | 110
Percentage of pts with g3+ hearing loss | 11 | 11

8. Secondary Outcome: Post-treatment Neurocognitive Function as Measured by the Estimated Full-scale IQ (FSIQ) by CSI Group Within Time Window 1 (4 - 15 Months Post Diagnosis).
Description: Post-treatment neurocognitive function was assessed. Full-scale IQ (FSIQ) is a representative measurement for neurocognitive function. FSIQ was measured by IQ tests. Assessments within the time window, from eligible and evaluable patients are reported. The time window is 4-15 months post diagnosis, only the assessments before progression date were reported. The Range of FSIQ is 50-150. A higher FSIQ is better.
Time Frame: 4 -15 months post diagnosis
Population: Only eligible & evaluable patients 3-7 years of age with FSIQ observations within time window were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 56 | 52
Scores on a scale | 93.8 (14.4) | 96.2 (15.0)

9. Secondary Outcome: Post-treatment Neurocognitive Function as Measured by the Estimated Full-scale IQ (FSIQ) by CSI Group Within Time Window 2 (27 - 48 Months Post Diagnosis)
Description: Post-treatment neurocognitive function was assessed. Full-scale IQ (FSIQ) is a representative measurement for neurocognitive function. FSIQ was measured by IQ tests. Assessments within the time window, from eligible and evaluable patients are reported. The time window is 27-48 months post diagnosis, only the assessments before progression date were reported. The range of FSIQ is 50 - 150. A higher FSIQ is better.
Time Frame: 27 - 48 months post diagnosis
Population: Only eligible & evaluable patients 3-7 years of age with FSIQ observations within time window were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 35 | 34
Scores on a scale | 92.2 (12.5) | 90.5 (13.3)

10. Secondary Outcome: Post-treatment Neurocognitive Function as Measured by the Estimated Full-scale IQ (FSIQ) by CSI Group Within Time Window 3 (49 - 72 Months Post Diagnosis)
Description: Post-treatment neurocognitive function was assessed. Full-scale IQ (FSIQ) is a representative measurement for neurocognitive function. FSIQ was measured by IQ tests. Assessments within the time window, from eligible and evaluable patients are reported. The time window is 49-72 months post diagnosis, only the assessments before progression date were reported. The Range of FSIQ is 50-150. A higher FSIQ is better.
Time Frame: 49 - 72 months post diagnosis
Population: Eligible and evaluable patients are reported.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 23 | 22
Scores on a scale | 90.5 (15.4) | 86.4 (13.5)

11. Secondary Outcome: Incidence of Grade 3+ Hearing Loss at 1-year Post Treatment as Assessed by CTCAE v4
Description: Proportions of patients with grade 3+ hearing impairment as assessed by CTCAE v4 at 1-year post treatment were calculated.
Time Frame: Up to 3 years
Population: Eligible & evaluable pts were included. Pts with anaplastic histology or disseminated/excess residual disease were not evaluable(NE). 26/23 IFRT/PFRT pts were NE, leaving 227 vs 237 eligible/evaluable pts. However some pts (28/22) weren't followed for at least 1-yr post-off tx (e.g., withdrew consent for FU or died), leaving 199 IFRT/215 PFRT pts.
Measure: Number; unit: Percentage of pts with g3+ hearing loss
Arm/Group | Involved Field Radiation (IFRT) | Posterior Fossa Radiation (PFRT)
Number analyzed (Participants) | 199 | 215
Percentage of pts with g3+ hearing loss | 8 | 8

12. Secondary Outcome: Incidence of Endocrine Dysfunction as Measured by Growth Hormone Stimulation Tests at the Time of Completion of Therapy by Radiotherapy (RT) Group
Description: Endocrine dysfunction was assessed by growth hormone stimulation (GHS) tests. We report the percentage of patients with abnormal growth hormone stimulation tests.
Time Frame: Post-treatment up to 3 years
Population: Only eligible & evaluable patients 3-7 years of age were included. Patients with anaplastic histology or disseminated/excess residual disease were not evaluable (NE). Availability of growth hormone stimulation test results were very limited. Only 3 out of 464 eligible and evaluable patients had this data available (2 PFRT patients and 1 IFRT).
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Involved Field Radiation (IFRT) | Posterior Fossa Radiation (PFRT)
Number analyzed (Participants) | 1 | 2
Percentage of patients | 0.0 [0.0 to 95.0] | 50.0 [2.5 to 97.5]

13. Secondary Outcome: Overall Survival (OS) by Molecular Subgroup Based on Methylation Arrays
Description: OS was defined as the time interval from date of study entry to date of death from any cause or to date of last contact for survivors. OS was estimated using the method of Kaplan and Meier. 3-year estimates are reported with 95% CI's.
Time Frame: 3 years
Population: 355 patients were classified into one of the medulloblastoma subgroups by methylation arrays and included in this analysis; 74 were Group 3 medulloblastoma, 154 were Group 4 medulloblastoma, 64 were SHH medulloblastoma, and 63 were WNT medulloblastoma patients.
Measure: Number (95% Confidence Interval); unit: Percent probability of overall survival
Groups:
- Group 3 Medulloblastoma: Includes eligible patients 3-21 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and classified as Group 3 medulloblastoma by methylation arrays
- Group 4 Medulloblastoma: Includes eligible patients 3-21 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and classified as Group 4 medulloblastoma by methylation arrays
- Sonic Hedgehog (SHH) Medulloblastoma: Includes eligible patients 3-21 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and classified as SHH medulloblastoma by methylation arrays
- Wingless (WNT) Medulloblastoma: Includes eligible patients 3-21 years of age without anaplastic histology or evidence of disseminated or ERD based on central review and classified as WNT medulloblastoma by methylation arrays
Arm/Group | Group 3 Medulloblastoma | Group 4 Medulloblastoma | Sonic Hedgehog (SHH) Medulloblastoma | Wingless (WNT) Medulloblastoma
Number analyzed (Participants) | 74 | 154 | 64 | 63
Percent probability of overall survival | 76.3 [66.5 to 86.1] | 97.3 [94.8 to 99.8] | 92.0 [85.1 to 98.9] | 98.3 [95.0 to 100.0]

14. Secondary Outcome: Progression-free Survival (PFS) by Molecular Subgroup Based on Methylation Arrays
Description: PFS was defined as the time interval from date of study entry to disease progression, relapse or death due to cancer or to last follow-up. Second malignancies and deaths from causes clearly not associated with tumor progression or recurrence were censored. PFS was estimated using the method of Kaplan and Meier. 3-year estimates are reported with 95% CI's.
Time Frame: 3 years
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage probability of PFS
Arm/Group | Group 3 Medulloblastoma | Group 4 Medulloblastoma | Sonic Hedgehog (SHH) Medulloblastoma | Wingless (WNT) Medulloblastoma
Number analyzed (Participants) | 74 | 154 | 64 | 63
Percentage probability of PFS | 70.6 [60.0 to 81.2] | 90.6 [85.9 to 95.3] | 90.4 [83.1 to 97.7] | 98.4 [95.3 to 100.0]

15. Secondary Outcome: Post-treatment Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) by CSI Group Within Time Window 1 (4-15 Months Post Diagnosis)
Description: Metacognition index (MI) was measured by BRIEF test. Assessments within the time window, from eligible and evaluable patients are reported. If the patient had disease progression, only the assessments before progression date were reported. The MI is a standard T- score, and it ranges from 0 to 100. The higher score reported suggests a higher level of dysfunction.
Time Frame: 4 - 15 months post diagnosis
Population: Only eligible & evaluable patients 3-7 years of age with MI values within time window were included.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 64 | 53
T-score | 50.7 (11.1) | 51.3 (9.6)

16. Secondary Outcome: Post-treatment Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) by CSI Group Within Time Window 2 (27-48 Months Post Diagnosis)
Description: as for outcome 15
Time Frame: 27-48 months post diagnosis
Population: Only eligible & evaluable patients 3-7 years of age with MI values within time window were included.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 27 | 27
T-score | 51.4 (10.6) | 55.0 (9.9)

17. Secondary Outcome: Post-treatment Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) by CSI Group Within Time Window 3 (49 - 72 Months Post Diagnosis)
Description: as for outcome 15
Time Frame: 49 - 72 months post diagnosis
Population: Only eligible & evaluable patients 3-7 years of age with MI values within time window were included.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Low-dose Craniospinal Radiation (LDSCI) | Standard-dose Craniospinal Radiation (SDCSI)
Number analyzed (Participants) | 21 | 22
T-score | 54.1 (10.7) | 58.6 (11.3)

18. Secondary Outcome: Compliance Rates for All Eligible and Evaluable Patients Enrolled Within Time Window 1 (4-15 Months Post Diagnosis)
Description: Compliance rates are calculated to monitor the compliance with long-term quality of life and functional status data submission. A patient will be compliant if the patient has metacognition index score. Compliance rates will be assessed at each of the 3 neurocognitive/quality of life assessment time windows. All eligible and evaluable patients enrolled will be used. Patients removed from treatment prior to the time of neuropsychological assessment (for reasons such as disease progression, death, withdrawal of consent, etc.) will not be included in the denominator to assess the compliance rate. The time window is 4 - 15 months post diagnosis.
Time Frame: 4-15 months post diagnosis
Population: All eligible and evaluable patients enrolled. Patients removed from treatment prior to the time of neuropsychological assessment (for reasons such as disease progression, death, withdrawal of consent, etc.) will not be included in the denominator to assess the compliance rate.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Eligible and Evaluable Patients: All eligible and evaluable patients enrolled on ACNS0331
Arm/Group | Eligible and Evaluable Patients
Number analyzed (Participants) | 448
Percentage of Participants | 58 [54 to 62]

19. Secondary Outcome: Compliance Rates for All Eligible and Evaluable Patients Enrolled Within Time Window 2 (27-48 Months Post Diagnosis)
Description: Compliance rates are calculated to monitor the compliance with long-term quality of life and functional status data submission. A patient will be compliant if the patient has metacognition index score. Compliance rates will be assessed at each of the 3 neurocognitive/quality of life assessment time windows. All eligible and evaluable patients enrolled will be used. Patients removed from treatment prior to the time of neuropsychological assessment (for reasons such as disease progression, death, withdrawal of consent, etc.) will not be included in the denominator to assess the compliance rate. The time window is 27 - 48 months post diagnosis.
Time Frame: 27-48 months post diagnosis
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eligible and Evaluable Patients
Number analyzed (Participants) | 395
Percentage of Participants | 32 [28 to 36]

20. Secondary Outcome: Compliance Rates for All Eligible and Evaluable Patients Enrolled Within Time Window 3 (49 - 72 Months Post Diagnosis)
Description: Compliance rates are calculated to monitor the compliance with long-term quality of life and functional status data submission. A patient will be compliant if the patient has metacognition index score. Compliance rates will be assessed at each of the 3 neurocognitive/quality of life assessment time windows. All eligible and evaluable patients enrolled will be used. Patients removed from treatment prior to the time of neuropsychological assessment (for reasons such as disease progression, death, withdrawal of consent, etc.) will not be included in the denominator to assess the compliance rate. The time window is 49 - 72 months post diagnosis.
Time Frame: 49 - 72 months post diagnosis
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eligible and Evaluable Patients
Number analyzed (Participants) | 131
Percentage of Participants | 69 [61 to 77]

ADVERSE EVENTS:
Description: All adverse events (grade 1 and higher) for all eligible patients (n=513) were included in this analysis. Serious AE's were based on whether an AdEERS report was filed OR whether the AE was a grade 5 AE (resulting in death). Of note, there was no other variable in the study database to indicate whether an AE was "serious" or not.
Arm/Group | Arm I (3-7 Years of Age, LDCSI, IFRT) | Arm II (3-7 Years of Age, LDCSI, PFRT) | Arm III (3-7 Years of Age, SDCSI, IFRT) | Arm IV (3-7 Years of Age, SDCSI, PFRT) | Arm V (8-21 Years of Age, SDCSI, IFRT) | Arm VI (8-21 Years of Age, SDCSI, PFRT)
Serious Adverse Events (participants affected / at risk) | 7/63 | 7/64 | 6/60 | 3/58 | 16/130 | 18/138
Other Adverse Events (participants affected / at risk) | 60/63 | 61/64 | 55/60 | 53/58 | 123/130 | 135/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (3-7 Years of Age, LDCSI, IFRT) (N=63) | Arm II (3-7 Years of Age, LDCSI, PFRT) (N=64) | Arm III (3-7 Years of Age, SDCSI, IFRT) (N=60) | Arm IV (3-7 Years of Age, SDCSI, PFRT) (N=58) | Arm V (8-21 Years of Age, SDCSI, IFRT) (N=130) | Arm VI (8-21 Years of Age, SDCSI, PFRT) (N=138)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalomyelitis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 4 (5) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (3-7 Years of Age, LDCSI, IFRT) (N=63) | Arm II (3-7 Years of Age, LDCSI, PFRT) (N=64) | Arm III (3-7 Years of Age, SDCSI, IFRT) (N=60) | Arm IV (3-7 Years of Age, SDCSI, PFRT) (N=58) | Arm V (8-21 Years of Age, SDCSI, IFRT) (N=130) | Arm VI (8-21 Years of Age, SDCSI, PFRT) (N=138)
Anemia (Blood and lymphatic system disorders) | 30 (109) | 30 (117) | 24 (125) | 27 (104) | 62 (278) | 55 (203)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (40) | 18 (32) | 22 (40) | 25 (48) | 42 (69) | 48 (68)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 8 (20) | 16 (27) | 12 (18) | 6 (11) | 16 (27) | 11 (23)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (7) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (10)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (8) | 2 (2) | 1 (2) | 1 (2) | 12 (22) | 13 (19)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (5) | 7 (15) | 4 (4) | 14 (19) | 21 (23)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (7) | 0 (0) | 8 (9) | 8 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (11) | 2 (2) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (8) | 5 (7) | 6 (9) | 4 (15) | 19 (34) | 14 (22)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (3) | 2 (2) | 5 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (8) | 3 (5) | 3 (4) | 2 (2) | 29 (56) | 22 (42)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8) | 4 (7) | 5 (8) | 9 (15) | 30 (49) | 31 (49)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 2 (4) | 2 (4) | 3 (4) | 12 (17) | 9 (21)
Fever (General disorders) | 4 (4) | 4 (5) | 6 (7) | 4 (5) | 9 (11) | 5 (6)
Gait disturbance (General disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (6) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 4 (5)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 2 (2)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 7 (9) | 4 (6) | 3 (3) | 6 (9) | 9 (9)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Encephalomyelitis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (2)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 12 (12) | 10 (16) | 15 (24) | 16 (35) | 28 (50) | 30 (48)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 5 (5)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 41 (148) | 36 (112) | 36 (145) | 37 (123) | 95 (415) | 95 (426)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 36 (113) | 35 (122) | 33 (96) | 32 (91) | 83 (302) | 87 (322)
Blood antidiuretic hormone abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 11 (18) | 7 (14) | 9 (19) | 6 (8) | 29 (65) | 21 (43)
Blood corticotrophin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 5 (8) | 10 (20) | 15 (30) | 6 (15) | 30 (76) | 30 (59)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Growth hormone abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Lymphocyte count decreased (Investigations) | 11 (60) | 14 (69) | 16 (97) | 9 (48) | 32 (220) | 38 (226)
Neutrophil count decreased (Investigations) | 58 (450) | 58 (421) | 51 (404) | 52 (362) | 118 (923) | 129 (932)
Platelet count decreased (Investigations) | 46 (253) | 43 (217) | 43 (269) | 41 (234) | 108 (687) | 118 (705)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (5) | 1 (1)
Weight loss (Investigations) | 8 (15) | 7 (20) | 8 (10) | 5 (6) | 24 (39) | 31 (43)
White blood cell decreased (Investigations) | 30 (147) | 22 (117) | 26 (136) | 25 (108) | 60 (322) | 63 (341)
Acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (2) | 3 (5) | 4 (10) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 15 (34) | 4 (13) | 9 (20) | 7 (16) | 33 (96) | 37 (109)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 5 (5) | 1 (1) | 11 (12) | 9 (12)
Hypercalcemia (Metabolism and nutrition disorders) | 10 (15) | 7 (9) | 13 (21) | 5 (6) | 18 (27) | 23 (44)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (14) | 3 (3) | 1 (2) | 2 (2) | 13 (24) | 8 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 3 (6) | 4 (7) | 9 (11) | 5 (8)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (4) | 2 (5) | 2 (3) | 0 (0) | 3 (7) | 4 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (9) | 1 (1) | 4 (10) | 2 (4) | 10 (11) | 5 (9)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 10 (21) | 11 (19) | 9 (14) | 9 (16) | 26 (49) | 20 (32)
Hypomagnesemia (Metabolism and nutrition disorders) | 20 (44) | 20 (51) | 29 (91) | 21 (41) | 54 (185) | 52 (157)
Hyponatremia (Metabolism and nutrition disorders) | 3 (8) | 0 (0) | 3 (5) | 3 (5) | 7 (11) | 5 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (8) | 1 (1) | 4 (10) | 1 (1) | 12 (19) | 10 (14)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 6 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (5) | 2 (9)
Growth suppression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 1 (3)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 5 (7) | 1 (2) | 1 (9) | 2 (7) | 2 (4) | 6 (20)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 4 (4) | 1 (2) | 8 (13) | 14 (23)
Hydrocephalus (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 2 (2)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Neuralgia (Nervous system disorders) | 7 (10) | 5 (16) | 16 (32) | 14 (20) | 35 (109) | 41 (95)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oculomotor nerve disorder (Nervous system disorders) | 1 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 35 (151) | 21 (84) | 34 (135) | 30 (124) | 92 (456) | 92 (431)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (90) | 17 (38) | 18 (70) | 14 (27) | 60 (221) | 65 (228)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (6)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 8 (10) | 9 (16)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 3 (3)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (5)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (3) | 3 (3) | 1 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (3) | 5 (6) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1) | 2 (3) | 1 (1) | 4 (12) | 3 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (4) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 4 (7)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No